CLINICAL TRIAL: NCT06485024
Title: Clinical Performance of Direct NanoHybrid Resin Composite Veneer Restorations Applied With or Without Modeling Resin:a Randomized Controlled Trial
Brief Title: Effect of Modeling Resin on Anterior Direct Composite Veneer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Azzazy ali, Master's student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MR in anterior
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Dental Wear; Dental Decay
MeSH Terms: conditions — Tooth Wear; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): the use of Modeling resin as the last layer applied to the NanoHybrid composite direct veneer
  Interventions: Device: Modeling Resin
- comparator (Active Comparator): the regular application of the NanoHybrid composite as a direct anterior veneer restoration
  Interventions: Device: Modeling Resin

INTERVENTIONS:
Device: Modeling Resin — it is the application of Modeling liquid to make easier manipulation and sculpting the composite veneer and reflect on its physical properties and clinical performance

SUMMARY:
the study will be conducted to evaluate the clinical performance of direct Nanohybrid resin composite veneer restorations applied with or without modeling resin

DETAILED DESCRIPTION:
ChatGPT This study aims to investigate the impact of modeling resin on the clinical performance of direct nanohybrid resin composite veneer restorations in anterior teeth. Resin composites are widely used in dental restorations due to their aesthetic qualities, but issues like discoloration and surface roughness can affect their longevity and patient satisfaction. Modeling resin, used to aid in composite placement and sculpting, has become common, but concerns exist regarding its effects on composite properties, particularly long-term color stability.

The research will employ a randomized controlled trial design with a two-arm parallel approach. Adult patients (18-45 years) with anterior tooth defects suitable for composite veneer restoration will be recruited. The intervention group will receive nanohybrid resin composite with modeling resin, while the comparator group will receive the composite without modeling resin. Outcomes will be assessed using modified USPHS criteria, including color stability, color match, anatomical form, marginal adaptation, marginal discoloration, retention rate, presence of secondary caries, and postoperative sensitivity, at baseline and at follow-up intervals of 1, 3, 6, and 12 months.

Statistical analysis will involve independent t-tests for intergroup comparisons and repeated measures ANOVA for intragroup comparisons, with a significance level set at 0.05. The study aims to determine if the use of modeling resin influences the clinical outcomes of resin composite veneer restorations. Ethics approval will be obtained, and confidentiality of participant data will be strictly maintained throughout the study period.

Overall, this research seeks to provide insights into optimizing the application of resin composites in dental practice to enhance patient outcomes and satisfaction

ELIGIBILITY:
Inclusion Criteria:

* • Adults (18-45Ys) with anterior tooth defects indicated for direct composite veneer restoration.

  * Males or females.
  * Community-dwelling
  * Have all his/her anterior teeth with sufficient enamel structure
  * With ≥ 1 anterior tooth defect
  * Have sufficient cognitive ability to understand consent procedures
  * Anterior tooth defect indicated for direct composite veneer
  * Vital upper or lower anterior teeth with no signs or symptoms of irreversible pulpitis.
  * Mobility grade: no clinical mobility
  * Plaque index ≤ 2

Exclusion Criteria:

* Patients younger than 18 or older than 45 years old • Disabilities.
* Systemic diseases or severe medically compromised.
* Lack of compliance.
* Evidence of severe bruxism, clenching or temporomandibular joint disorders.
* Cognitive impairment

Periapical pathosis or signs of pulpal pathology.

* Malocclusion
* Possible prosthodontic restoration within 1 year.
* Non-vital tooth.
* Endodontically treated tooth.
* Severe periodontal affection or tooth indicated for extraction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
comparison of Color stability with and without the intervention | baseline and after one year
  by using Spectrophotometer to measure the color considering the intervention

SECONDARY OUTCOMES:
comparing the effect of the intervention on color match | baseline and after one year
  using the modefied USPHS criteria
comparing the effect of the intervention on anatomical form | baseline and after one year
  using the modefied USPHS criteria
comparing the effect of the intervention on surface texture | baseline and after one year
  using the modefied USPHS criteria
comparing the effect of the intervention on marginal adaptation | baseline and after one year
  using the modefied USPHS criteria
comparing the effect of the intervention on marginal discoloration | baseline and after one year
  using the modefied USPHS criteria
comparing the effect of the intervention on retention rate | baseline and after one year
  using the modefied USPHS criteria
comparing the effect of the intervention on postoperative sensitivity | baseline and after one year
  using the modefied USPHS criteria
comparing the effect of the intervention on recurrent caries | baseline and after one year
  using the modefied USPHS criteria

REFERENCES:
- [Background] Munchow EA, Sedrez-Porto JA, Piva E, Pereira-Cenci T, Cenci MS. Use of dental adhesives as modeler liquid of resin composites. Dent Mater. 2016 Apr;32(4):570-7. doi: 10.1016/j.dental.2016.01.002. Epub 2016 Feb 3. PMID 26850844
- [Background] Stefanski S, van Dijken JW. Clinical performance of a nanofilled resin composite with and without an intermediary layer of flowable composite: a 2-year evaluation. Clin Oral Investig. 2012 Feb;16(1):147-53. doi: 10.1007/s00784-010-0485-8. Epub 2010 Nov 23. PMID 21104100
- [Result] Rosentritt M, Esch J, Behr M, Leibrock A, Handel G. In vivo color stability of resin composite veneers and acrylic resin teeth in removable partial dentures. Quintessence Int. 1998 Aug;29(8):517-22. PMID 9807133
- [Result] Al-Asmar AA, Ha Sabrah A, Abd-Raheam IM, Ismail NH, Oweis YG. Clinical evaluation of reasons for replacement of amalgam vs composite posterior restorations. Saudi Dent J. 2023 Mar;35(3):275-281. doi: 10.1016/j.sdentj.2023.02.003. Epub 2023 Mar 4. PMID 37091274
- [Result] Bhadra D, Shah NC, Kishan KV, Dedania MS. An in vitro comparative evaluation of commonly consumed catechu and catechu with lime on surface roughness and color stability of the conventional nano-hybrid composite. J Conserv Dent. 2019 Jan-Feb;22(1):87-91. doi: 10.4103/JCD.JCD_181_18. PMID 30820089
- [Result] Crins LAMJ, Opdam NJM, Kreulen CM, Bronkhorst EM, Sterenborg BAMM, Huysmans MCDNJM, Loomans BAC. Randomized controlled trial on the performance of direct and indirect composite restorations in patients with severe tooth wear. Dent Mater. 2021 Nov;37(11):1645-1654. doi: 10.1016/j.dental.2021.08.018. Epub 2021 Sep 6. PMID 34497023
- [Result] Demarco FF, Collares K, Correa MB, Cenci MS, Moraes RR, Opdam NJ. Should my composite restorations last forever? Why are they failing? Braz Oral Res. 2017 Aug 28;31(suppl 1):e56. doi: 10.1590/1807-3107BOR-2017.vol31.0056. PMID 28902236
- [Result] Cortopassi LS, Shimokawa CAK, Willers AE, Sobral MAP. Surface roughness and color stability of surface sealants and adhesive systems applied over a resin-based composite. J Esthet Restor Dent. 2020 Jan;32(1):64-72. doi: 10.1111/jerd.12548. Epub 2019 Nov 18. PMID 31737981
- [Result] Malekipour MR, Sharafi A, Kazemi S, Khazaei S, Shirani F. Comparison of color stability of a composite resin in different color media. Dent Res J (Isfahan). 2012 Jul;9(4):441-6. PMID 23162586
- [Result] Gianordoli-Neto R, Padovani GC, Mondelli J, de Lima Navarro MF, Mendonca JS, Santiago SL. Two-year clinical evaluation of resin composite in posterior teeth: A randomized controlled study. J Conserv Dent. 2016 Jul-Aug;19(4):306-10. doi: 10.4103/0972-0707.186446. PMID 27563176
- [Result] Heintze SD, Rousson V, Hickel R. Clinical effectiveness of direct anterior restorations--a meta-analysis. Dent Mater. 2015 May;31(5):481-95. doi: 10.1016/j.dental.2015.01.015. Epub 2015 Mar 13. PMID 25773188
- [Result] Maia TS, Lima TD, Ramos VM, Faria-E-Silva AL, Menezes MS. Effect of modeling liquids on resin composite roughness and color parameters after staining and toothbrushing. Braz Oral Res. 2023 Mar 31;37:e024. doi: 10.1590/1807-3107bor-2023.vol37.0024. eCollection 2023. PMID 37018806
- [Result] Paolone G, Mazzitelli C, Josic U, Scotti N, Gherlone E, Cantatore G, Breschi L. Modeling Liquids and Resin-Based Dental Composite Materials-A Scoping Review. Materials (Basel). 2022 May 24;15(11):3759. doi: 10.3390/ma15113759. PMID 35683057
- [Result] Pizzolotto L, Moraes RR. Resin Composites in Posterior Teeth: Clinical Performance and Direct Restorative Techniques. Dent J (Basel). 2022 Nov 27;10(12):222. doi: 10.3390/dj10120222. PMID 36547038
- [Result] Cetin AR, Unlu N. One-year clinical evaluation of direct nanofilled and indirect composite restorations in posterior teeth. Dent Mater J. 2009 Sep;28(5):620-6. doi: 10.4012/dmj.28.620. PMID 19822994
- [Result] Sedrez-Porto JA, Munchow EA, Brondani LP, Cenci MS, Pereira-Cenci T. Effects of modeling liquid/resin and polishing on the color change of resin composite. Braz Oral Res. 2016 Aug 18;30(1):S1806-83242016000100275. doi: 10.1590/1807-3107BOR-2016.vol30.0088. PMID 27556554